CLINICAL TRIAL: NCT02330939
Title: Impact of Fats And Carbohydrates Quality on Postprandial glycemIc Response in People With Type 1 diabEtes on Insulin Pump (FACILE Study)
Brief Title: Fats And Carbohydrates Quality on Postprandial glycemIc Response in Type 1 Diabetes
Acronym: FACILE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, rivellese angela, professor, Federico II University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 980/14
Record Dates: First submitted 2015-01-01; First posted 2015-01-05 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2015-01

CONDITIONS: Type 1 Diabetes
Keywords: Postprandial glycemia; Momounsaturated fatty acids; Saturated fatty acids; Glycemic index; Glycemic load; Sensor augmented pump system
MeSH Terms: conditions — Diabetes Mellitus, Type 1

ARMS (6):
- Low fat- Low glycemic index (Active Comparator): Participants consumed a meal with low glycemic index and poor in fat
  Interventions: Other: Low fat- Low glycemic index meal
- MUFA- Low glycemic index (Experimental): Participants consumed a meal with low glycemic index and rich in MUFA
  Interventions: Other: MUFA- Low glycemic index meal
- SAFA- Low glycemic index (Experimental): Participants consumed a meal with low glycemic index and rich in SAFA
  Interventions: Other: SAFA- Low glycemic index meal
- Low fat- High glycemic index (Active Comparator): Participants consumed a meal with high glycemic index and low in fat
  Interventions: Other: Low fat- High glycemic index meal
- MUFA- High glycemic index (Experimental): Participants consumed a meal with high glycemic index and rich in MUFA
  Interventions: Other: MUFA- High glycemic index meal
- SAFA- High glycemic index (Experimental): Participants consumed a meal with high glycemic index and rich in SAFA
  Interventions: Other: SAFA- High glycemic index meal

INTERVENTIONS:
Other: Low fat- Low glycemic index meal
  Arms: Low fat- Low glycemic index
Other: MUFA- Low glycemic index meal
  Arms: MUFA- Low glycemic index
Other: SAFA- Low glycemic index meal
  Arms: SAFA- Low glycemic index
Other: Low fat- High glycemic index meal
  Arms: Low fat- High glycemic index
Other: MUFA- High glycemic index meal
  Arms: MUFA- High glycemic index
Other: SAFA- High glycemic index meal
  Arms: SAFA- High glycemic index

SUMMARY:
The purpose of this study is to determine whether dietary fats may affect postprandial glycemic response differently according to their quality, and these effects may differ whether they are assumed in the context of meals with high or low glycemic index in patients with type 1 diabetes. This interaction between quality of fat and glycemic index of carbohydrates may have clinical implication for the calculation of prandial insulin dose in these patients.

ELIGIBILITY:
Inclusion Criteria:

-Type 1 diabetes treated by insulin pump

Exclusion Criteria:

* Pregnancy
* Celiac disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
postprandial incremental glucose AUC | 6 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Medicine and Surgery, Naples, Italy

REFERENCES:
- [Derived] Bozzetto L, Alderisio A, Clemente G, Giorgini M, Barone F, Griffo E, Costabile G, Vetrani C, Cipriano P, Giacco A, Riccardi G, Rivellese AA, Annuzzi G. Gastrointestinal effects of extra-virgin olive oil associated with lower postprandial glycemia in type 1 diabetes. Clin Nutr. 2019 Dec;38(6):2645-2651. doi: 10.1016/j.clnu.2018.11.015. Epub 2018 Dec 4. PMID 30567626
- [Derived] Bozzetto L, Alderisio A, Giorgini M, Barone F, Giacco A, Riccardi G, Rivellese AA, Annuzzi G. Extra-Virgin Olive Oil Reduces Glycemic Response to a High-Glycemic Index Meal in Patients With Type 1 Diabetes: A Randomized Controlled Trial. Diabetes Care. 2016 Apr;39(4):518-24. doi: 10.2337/dc15-2189. Epub 2016 Feb 9. PMID 26861923